CLINICAL TRIAL: NCT00061373
Title: Combination Anti-Platelet and Anti-Coagulation Treatment After Lysis of Ischemic Stroke Trial (CATALIST)
Acronym: CATALIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030171; 03-N-0171
Record Dates: First submitted 2003-05-23; First posted 2003-05-26 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2012-12

CONDITIONS: Ischemic Stroke
Keywords: Alteplase; Recombinant tissue plasminogen activator; Reperfusion therapy; Magnetic Resonance Imaging; Clinical Trial; Tinzaparin; Eptifibatide; Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Tinzaparin; Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI Selected Patients (Experimental): Patients are eligible for the MRI arm if all clinical and all MRI inclusion and exclusion criteria are met.
  A single dose of aspirin 81 mg orally (or rectal dose equivalent), a single weight-based dose of subcutaneous tinzaparin sodium. Possible dose escalated iv eptifibatide.
  Interventions: Drug: Aspirin; Drug: tinzaparin sodium; Drug: eptifibatide
- non-MRI Selected Patients (Experimental): Patients are eligible for the non-MRI arm if all clinical inclusion-exclusion criteria are met, if MRI is contraindicated or if MRI compromises iv tPA delivery within 3-hours of symptom onset.
  A single dose of aspirin 81 mg orally (or rectal dose equivalent) and a single weight-based dose of subcutaneous tinzaparin sodium. Possible dose escalated iv eptifibatide.
  --------------------------------------------------------------------------------
  Interventions: Drug: Aspirin; Drug: tinzaparin sodium; Drug: eptifibatide

INTERVENTIONS:
Drug: Aspirin — A single 81 mg aspirin tablet orally (or rectal suppository equivalent dose) given as soon as possible after start of standard iv tPA and consent.
Drug: tinzaparin sodium — A single weight-based dose of 80 anti-Xa International Units/kilogram (IU/kg)administered by subcutaneous (SQ) injection.
  Other Names: Innohep (registered trademark)
Drug: eptifibatide — Eptifibatide administered iv according to dose escalation group. The five dosing groups for eptifibatide are 0, 45 µg/kg bolus, 90 µg/kg bolus, 90 µg/kg bolus plus 0.25 µg/kg/min infusion for 24 hours, and 90 µg/kg bolus plus 0.5 µg/kg/min infusion for 24 hours.
  Other Names: Integrilin (registered trademark)

SUMMARY:
Ischemic stroke is caused by a blood clot that blocks the flow of blood to the brain and damages brain cells. The clot, or thrombus, is made up of platelets and fibrin. The medicine alteplase, also known as tPA , is the standard drug used to treat patients with acute ischemic stroke. tPA attacks the fibrin portion of the blood clot. While intravenous (iv) tPA alone is effective in treating the fibrin part of the clot approximately 30% of the time, adding other commercially available drugs such eptifibatide to treat other clot components may improve the effectiveness of iv tPA therapy.

This is a clinical trial to determine an acceptable dose of eptifibatide in combination with aspirin, the low molecular weight heparin tinzaparin, and standard iv tPA therapy for the treatment of acute ischemic stroke. Use of clinical and imaging based selection criteria are hypothesized to contribute to treatment safety by selecting patients at lower risk of intracerebral hemorrhage. Also,selection and evaluation of patients by magnetic resonance imaging (MRI) criteria will result in a different risk to benefit ratio than selecting patients without MRI criteria and will lead to a different acceptable dose.

DETAILED DESCRIPTION:
Study Population: All acute ischemic stroke patients treated with standard iv tPA therapy within 3 hours from stroke onset will be considered for study participation. Patient will be selected by criteria to minimize likelihood of toxicity and maximize likelihood of response. These criteria include age 18-85 years old acute ischemic stroke of moderate severity measured using the National Institutes of Health Stroke Scale Stroke Scale (NIHSS) less than 22 for left hemisphere strokes, less than 17 for others) and no other clinical, radiological or laboratory features associated with increased risk of hemorrhage of thrombolytic therapy. In the MRI arm of the trial, patients must have positive MRI evidence of hypoperfusion corresponding to the acute stroke symptoms and no MRI evidence of chronic micro-hemorrhages.

Design: This is an open-label, dose escalation, safety and proof of principle clinical trial. All patients will receive iv tPA therapy plus 81 mg aspirin orally (or 150 mg rectally) and 80 anti Xa IU/kg tinzaparin subcutaneously and some patients will receive iv eptifibatide. Intravenous eptifibatide will be given in a dose-escalating manner. The five dosing groups for eptifibatide are 0, 45 micro g/kg bolus, 90 micro g/kg bolus, 90 micro g/kg bolus plus 0.25 micro g/kg/min infusion for 24 hours, and 90 mg/kg bolus plus 0.5 micro g/kg/min infusion for 24 hours. Investigational therapy is to begin as early as possible but no later than 6 hours after the onset of the patient's symptoms. Two arms - an MRI and a non-MRI arm - will receive identical drug regimes,and dose escalation will proceed independently in either arm.

A maximum of 100 patients in each arm will be studied, a minimum of 15 patients treated at each dose level. The outcomes will be monitored by a Data and Safety Monitoring Board (DSMB). The DSMB will have the authority to stop or recommend modifications of the trial for safety concerns throughout the trial and after any occurrence of severe adverse events (SAE). Dose escalation from one dose level to the next will be contingent on DSMB approval.

Outcome Measures: The primary safety endpoint for determination of toxicity will be any one of the following: symptomatic intracranial hemorrhage (ICH), major systemic hemorrhage, or other SAE related to study drug administration, within 72 hours from start of therapy. Adverse events will be monitored for 30 days. The primary efficacy endpoint for response in the MRI arm will be reperfusion as measured by perfusion weighted imaging (PWI) at both 2 hours and 24 hours after start of therapy and substantial clinical recovery at 24 hours for the non-MRI arm. Clinical outcome variables and imaging variables will be recorded and analyzed in secondary and exploratory analyses. If an acceptable dose of eptifibatide is identified, that dose of eptifibatide will be investigated in a subsequent randomized placebo-controlled trial.

MRI and CT are used as radiological measures of brain hemorrhage. The NIH Stroke Scale (NIHSS) is used to measure neurological worsening or recovery.

The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute stroke on the levels of consciousness, language, neglect, visual-field loss, extra ocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patient's ability to answer questions and perform activities. Ratings for each of the 15 items are scored. Patients who have a score of 0 are considered to have "normal" examination. Patients with a score of 40 have the most severe stroke symptoms.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Diagnosis of acute ischemic stroke with planned start of intravenous tPA. Acute ischemic stroke is defined as a measurable neurological deficit of sudden onset, presumed secondary to focal cerebral ischemia. Stroke onset will be defined as the time the patient was last known to be without the new clinical deficit. If the stroke started during sleep, stroke onset will be recorded as the time the patient was last known to be at baseline.
2. Disabling neurological deficit attributable to acute ischemic stroke.
3. NIHSS less than or equal to 21 for left hemisphere strokes, NIHSS less than or equal to 16 for others.
4. Age 18-85 years, inclusive.
5. Body weight greater than 50 kg.

   For MRI Arm only:
6. Screening MRI diagnostic of focal cerebral ischemia corresponding to the clinical deficits. The MRI evaluation must involve echo planar diffusion weighted imaging, magnetic resonance angiography(MRA),and MRI perfusion. A normal appearing MRA with an appropriate perfusion deficit is eligible. An apparent stenosis or occlusion on MRA with normal appearing perfusion distally will not be eligible. Poor quality or uninterpretable MRA will not make patient ineligible. Patients who have a normal appearing diffusion weighted image (DWI) are eligible.
7. Evidence on perfusion weighted image (PWI) MRI or a perfusion defect corresponding to the acute stroke syndrome. The PWI will be assessed by relative mean transit time (MTT) images obtained prior to the start of tPA therapy.

EXCLUSION CRITERIA:

1. Current participation in another study with an investigational drug or device within, prior participation in the present study, or planned participation in another therapeutic trial, prior to the final (day 30) assessment in this trial.
2. Symptoms suggestive of subarachnoid hemorrhage, even if CT or MRI scan is negative for hemorrhage.
3. Evidence of acute myocardial infarction defined as having at least two of the following three features: 1) Chest pain suggestive of cardiac ischemia; 2) EKG findings of ST elevation of more greater than 0.2 millivolts (mV) in 2 contiguous leads, new onset left bundle branch block, ST segment depression, or T-wave inversion; 3) Elevated troponin I.
4. Acute Pericarditis.
5. Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.
6. Patients who would refuse blood transfusions if medically indicated.
7. Neurological deficit that has led to stupor or coma (NIHSS level of consciousness [item I a] score greater than or equal to 2).
8. High clinical suspicion of septic embolus.
9. Minor stroke with non-disabling deficit or rapidly improving neurological symptoms.
10. Baseline NIHSS greater than 21 for left hemisphere stroke or greater than 16 for others.
11. Evidence of acute or chronic ICH by head CT or MRI.
12. CT or MRI evidence of non-vascular cause for the neurological symptoms.
13. Signs of mass effect causing shift of midline structures on CT or MRI.
14. Persistent hypertension with systolic BP greater than 185 mmHg or diastolic BP greater than 110 mmHg (mean of 3 consecutive arm cuff readings over 20-30 minutes), not controlled by antihypertensive therapy or requiring nitroprusside for control.
15. Anticipated need for major surgery within 72 hours after start of study drugs, such as a carotid endarterectomy or hip fracture repair.
16. Any intracranial surgery, intraspinal surgery, or serious head trauma (any head injury that required hospitalization) within the past 3 months.
17. Stroke within the past 3 months.
18. History of ICH at any time in the past.
19. Major trauma at the time of stroke, such as a hip fracture.
20. Blood glucose greater than 200 milligrams per diluent (mg/dl).
21. Presence or history of intracranial neoplasm (except small meningiomas) or arteriovenous malformation.
22. Intracranial aneurysm, unless surgically or endovascularly treated more than 3 months before.
23. Seizure at the onset of stroke.
24. Active internal bleeding.
25. Major hemorrhage (requiring transfusion, surgery or hospitalization) in the past 21 days.
26. Major surgery, serious trauma, lumbar puncture, arterial puncture at a non-compressible site, or biopsy of a parenchymal organ in last 14 days. Major surgical procedures include but are not limited to the following: major thoracic or abdominopelvic surgery, neurosurgery, major limb surgery, carotid endarterectomy or other vascular surgery, and organ transplantation. For non-listed procedures, the operating surgeon should be consulted to assess the risk.
27. Presumed or documented history of vasculitis.
28. Known systemic bleeding or platelet disorder, e.g., von Willebrand's disease, hemophilia, idiopathic thrombocytopenia purpura (ITP),thrombotic thrombocytopenic purpura (TTP), others.
29. History of heparin induced thrombocytopenia.
30. Platelet count less than 100,000 cells/microliter.
31. Congenital or acquired coagulopathy (e.g. , secondary to anticoagulants) causing either of the following:

    1. Activated partial thromboplastin time (aPTT) prolongation greater than 2 seconds above the upper limit of normal for local laboratory, except if due to isolated factor twelve (XII) deficiency.
    2. International normalized ratio (INR) greater than or equal to 1.4. Patients receiving warfarin prior to entry are eligible provided INR is less than 1.4 and warfarin can be safely discontinued for at least 48 hours.
32. Life expectancy less than 3 months.
33. Other serious illness, e.g., severe hepatic, cardiac, or renal failure; acute myocardial infarction; or complex disease that may confound treatment assessment.
34. Severe renal failure: Serum creatinine greater than 4.0 mg/dL or dependency on renal dialysis.
35. Aspartate aminotransferase (AST) or Alanine transaminase(ALT) greater than 3 times the upper limit of normal for the local laboratory.
36. Treatment of the qualifying stroke with any thrombolytic, anti-thrombotic or glycoprotein inhibitor(GPIIbIIIa)outside of this protocol.
37. Any administration of a thrombolytic drug in the prior 7 days.
38. Treatment of the qualifying stroke with intravenous heparin unless aPTT prolongation is no greater than 2 seconds above the upper limit of normal for local laboratory prior to study drug initiation.
39. Treatment of the qualifying stroke with a low molecular weight heparin or heparinoid.
40. Known hypersensitivity to alteplase, aspirin, tinzaparin, eptifibatide, heparin, sulfites, benzyl alcohol, or pork products.
41. Anticoagulation (evidenced by abnormal INR, aPTT, or platelet count) caused by herbal therapy.
42. Known history of alcohol or illicit drug use (e.g. prior to study drug administration)

    FOR non-MRI arm only (items 43-44):
43. Ischemic changes on screening CT of greater than approximately one third of the territory of the middle cerebral artery territory by qualitative assessment.
44. Patients who were excluded by screening MRI, except for exclusions item 45 (contraindication to MRI) and item 46 (PWI was not obtained or is uninterpretable) and item 51 (MRI not obtainable because it would have put the patient out of the 3 hour time window for tPA).

    FOR MRI arm only (items 45-51):
45. Contraindication to MRI scan.
46. PWI not obtained or uninterpretable.
47. No MTT defect corresponding to acute stroke deficit.
48. Satellite DWI hyperintensity with corresponding hyperintensity on T2 weighted image or FLAIR in a vascular territory different than the index stroke
49. DWI abnormality larger than approximately one third of the territory of the middle cerebral artery territory by qualitative assessment.
50. Evidence of multiple microbleeds on gradient echo MRI (GRE).
51. Patient has a contraindication to gadolinium contrast agent: prior adverse reaction to gadolinium or estimated glomerular filtration rate(GFR) less than 60 milliliters per minute (mL/min).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-05; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Warach, MD, PhD, Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (3):
- United States (3):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Suburban Hospital, Bethesda, Maryland

REFERENCES:
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Background] Albers GW, Bates VE, Clark WM, Bell R, Verro P, Hamilton SA. Intravenous tissue-type plasminogen activator for treatment of acute stroke: the Standard Treatment with Alteplase to Reverse Stroke (STARS) study. JAMA. 2000 Mar 1;283(9):1145-50. doi: 10.1001/jama.283.9.1145. PMID 10703776
- [Background] Califf RM. Combination therapy for acute myocardial infarction: fibrinolytic therapy and glycoprotein IIb/IIIa inhibition. Am Heart J. 2000 Feb;139(2 Pt 2):S33-7. doi: 10.1067/mhj.2000.104090. PMID 10650314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this clinical trial opened in 2004 and closed in 2009. Patients who presented to one of two metropolitan Washington, DC hospitals with acute ischemic stroke and who treated with standard iv tPA were screened for study enrollment.
Pre-assignment Details: Enrollment into the MRI was preferential. If patients had contraindications to MRI or acquisition of MRI delayed treatment with iv tPA, they were enrolled in the non-MRI arm of the study.
Groups:
- MRI- Selected Patients: Patients eligible for the MRI arm met all clinical and MRI inclusion and exclusion criteria.
  Patients received a single dose of aspirin 81 mg orally (or rectal dose equivalent)and a single SQ dose of tinzaparin sodium, 80 anti-Xa IU/kg as soon after iv tPA and consent but within 6 hours of the start of iv tPA.
- Non-MRI Selected Patients: Patients eligible for the non-MRI arm met all clinical inclusion-exclusion criteria, had MRI is contraindications or the acquisition of MRI would have compromised iv tPA delivery within the standard treatment window.
  Patients received a single dose of aspirin 81 mg orally (or rectal dose equivalent)and a single SQ dose of tinzaparin sodium, 80 anti-Xa IU/kg as soon after iv tPA and consent but within 6 hours of the start of iv tPA.
Period: Overall Study
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Started | 15 | 3
Aspirin and Tinzaparin | 15 | 3
Completed | 15 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients | Total
Number analyzed (Participants) | 15 | 3 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 10 | 1 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 59 (7) | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 15 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Intracerebral Hemorrhage (ICH)
Description: This is a primary safety outcome or toxicity measure for all subjects.
  Symptomatic ICH is defined as the presence of two conditions: evidence of hemorrhage on the 72-hour head CT and an increase in the NIHSS score of 4 or more points from the prior examination. Hemorrhage classifications are according to European Cooperative Acute Stroke Study (ECASS).
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute stroke on the levels of consciousness, language, neglect, visual-field loss, extra ocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patient's ability to answer questions and perform activities. Ratings for each of the 15 items are scored. Patients who have a score of 0 are considered to have "normal" examination. Patients with a score of 40 have the most severe stroke symptoms.
Time Frame: From the start of study drugs and prior to the 72-hour safety head CT
Population: All patients had a 72-hour safety head CT performed
Measure: Number; unit: participants
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Number analyzed (Participants) | 15 | 3
participants | 1 | 1

2. Primary Outcome: Major Systemic Hemorrhage
Description: Major systemic hemorrhage is defined bleeding associated with an adjusted decrease in hemoglobin of greater than 5 grams per diluent (g/dL), or and adjusted decrease in hematocrit greater than or equal to 15 percentage points or bleeding causing persistent or significant disability or incapacity such as hemorrhage in the eye.
Time Frame: From the start of study drugs and prior to 72-hour head CT
Population: All patients completed 72-hour safety evaluation
Measure: Number; unit: participants
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Number analyzed (Participants) | 15 | 3
participants | 0 | 0

3. Primary Outcome: Other Serious Adverse Event Related to Study Drug Administration, Including Death.
Description: This is a primary safety outcome for all subjects.
Time Frame: From start of study drugs and prior to 72-hour head CT
Population: All Patients completed 72-hour study safety evaluation
Measure: Number; unit: participants
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Number analyzed (Participants) | 15 | 3
participants | 0 | 0

4. Primary Outcome: MRI Selected Arm: Complete Brain Reperfusion
Description: This is the primary response outcome measure for patients in the MRI arm. A positive response is measured by evidence of complete reperfusion (or restoration of blood flow)on the perfusion weighted images (PWI) and mean transit time (MTT) maps of MRIs at 2 hours and sustained at 24 hours.
Time Frame: up to 24 hours from the start of study drugs
Population: Complete reperfusion at 2 and 24 hours was measured in MRI-selected patients only.
Measure: Number; unit: participants
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Number analyzed (Participants) | 14 | 0
participants | 0 |

5. Primary Outcome: Non-MRI Selected Arm: Substantial Clinical Recovery (Non-MRI Arm)
Description: This is the primary response outcome measure for subjects in the non-MRI arm. A positive response is measured by a 7 point or more improvement in the NIHSS or for those with less than 7 points at baseline,complete resolution of stroke symptoms.
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute stroke on the levels of consciousness, language, neglect, visual-field loss, extra ocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patient's ability to answer questions and perform activities. Ratings for each of the 15 items are scored. Patients who have a score of 0 are considered to have "normal" examination. Patients with a score of 40 have the most severe stroke symptoms.
Time Frame: up to 24 hours from the start of study drugs
Population: Clinical improvement on NIHSS of 7 points or greater at 72 hours is the primary response outcome for non-MRI selected patients. Clinical response outcome was analyzed on all patients enrolled; MRI selected and non-selected patients.
Measure: Number; unit: participants
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Number analyzed (Participants) | 15 | 3
participants | 3 | 2

6. Secondary Outcome: Bleeding Events
Description: Bleeding events of any type, severity and at any time throughout the 30-day trial period.
Time Frame: 2 hr, 24 hr, 72 hr, 5 days, 30 days from start of study drugs
Population: All bleeding events that occurred among all patients enrolled and throughout the 30-day trial period but not classified as a primary outcome event. Bleeding events in this category include asymptomatic ICH(aICH);major systemic bleeding after 72 hours or minor and non-significant bleeding at anytime within the 30-day period.
Measure: Number; unit: participants
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Number analyzed (Participants) | 15 | 3
participants | 8 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start of study drug administration through the 30-day study period.
Description: All cases of ICH were reported to and reviewed by the DSMB. Patients with symptomatic ICH prior to the 72-hour head CT were reviewed by the DSMB prior to enrollment of new patients.
Arm/Group | MRI- Selected Patients | Non-MRI Selected Patients
Serious Adverse Events (participants affected / at risk) | 4/15 | 2/3
Other Adverse Events (participants affected / at risk) | 12/15 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI- Selected Patients (N=15) | Non-MRI Selected Patients (N=3)
Neurological Worsening (Nervous system disorders) | 1 (1) | 0 (0) — measured by change in NIHSS score of 4 or more points
Symptomatic ICH (Nervous system disorders) | 1 (1) | 1 (1) — reading of non-contrast head CT for all and reading of gradient echo (GRE) for MRI-selected patients
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 2 (2) — doppler confirmed
Non-ST Segment Elevation Myocardial Infarction (NSTEMI) (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Systemic Bleeding/Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Metabolic Disturbance (Endocrine disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI- Selected Patients (N=15) | Non-MRI Selected Patients (N=3)
Fever (Infections and infestations) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Metabolic Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Pain, lower extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus bradycardia, asymptomatic (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 2 (3) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Asymptomatic ICH (Nervous system disorders) | 6 (6) | 1 (1)
Ischemic Stroke, New (Nervous system disorders) | 1 (1) | 0 (0)
Expansion of ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Mood Alteration (Nervous system disorders) | 1 (1) | 0 (0)
Neurological Worsening (Nervous system disorders) | 2 (2) | 0 (0)
Labored Breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
All patients enrolled were dosed with aspirin and tinzaparin. None of the patients received iv eptifibatide. The study was closed prior to dosing with eptifibatide due to slow recruitment over the 5-year trial period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes